CLINICAL TRIAL: NCT04376294
Title: Using of Extracorporeal Shockwave Therapy in Treatment Of Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Prof.Dr. Emad Samuel Boles Saweeres (Unknown); Prof.Dr Nadia Abdelazim fayaz (Unknown); Mr.Mohamed Nasser Kise Helmy (Unknown)
Responsible Party: Principal Investigator, Nasr Awad Abdelkader Othman, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002042
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Achilles Tendinopathy
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): This group received Extracorporeal Shockwave Therapy(ESWT) + conservative Physical Therapy Treatment (eccentric training + stretching exercise)
  Interventions: Device: Extracorporeal Shockwave Therapy(ESWT); Other: Eccentric training of the calf muscle:; Other: Gastrocnemius, soleus, and hamstring stretch
- Control group (Active Comparator): This group received conservative physical therapy treatment(eccentric training + stretching exercise) only.
  Interventions: Other: Eccentric training of the calf muscle:; Other: Gastrocnemius, soleus, and hamstring stretch

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy(ESWT) — Each session of Extracorporeal Shockwave Therapy(ESWT) consists of 2000 pulses with a pressure of 3 bars (equals an energy flux density of 0.1 mJ/mm²), and treatment frequency of 8 pulses/sec
  Arms: Study group
Other: Eccentric training of the calf muscle: — The patients were asked to stand with all their body weight on the injured leg on a wooden step. From an upright body position and standing with all body weight on the forefoot, with the ankle joint in plantar flexion. The calf muscle is loaded by having the patient lower the affected limb down by dorsiflexion the ankle until the plantar aspect of the heel lay below the level of the step, and the ankle is in maximum dorsiflexion.
Other: Gastrocnemius, soleus, and hamstring stretch — Stretching every muscle for 30 seconds. Each stretch was performed 3 times (holding for 30 seconds and rest for 30 seconds). All these stretches were performed directly after the eccentric exercises twice/day for 7 days/week for weeks

SUMMARY:
The purpose of this study was to determine the effect of extracorporeal Shock wave therapy (ESWT) on functional activity and pain in patients with Achilles tendinopathy

DETAILED DESCRIPTION:
Fifty patients of both sexes with Achilles tendinopathy aged 18-40 years, were assigned randomly into two equal groups. The study group received ESWT in addition to a conservative physical therapy program for four weeks, while the control group received a conservative physical therapy program only. Pain and functional mobility were assessed before and after treatment through a visual analog scale (VAS) and Victorian Institute of sports assessment - Achilles questionnaire (VISA-A), respectively

ELIGIBILITY:
Inclusion criteria

* Clinical history of Achilles tendon pain for at least six months
* A minimum of three months conservative treatment administered without benefit for at least four weeks before ESWT.

Exclusion Criteria:

* Patients underwent physical therapy in the four weeks prior enrollment to study.
* Patients had taken non-steroidal anti-inflammatory medication during the previous week
* Patients had received peritendinous injections of a local anesthetic or corticosteroid within last 4 weeks
* Patients had bilateral Achilles tendinopathy
* Patients with other conditions that could significantly contribute to posterior ankle pain (osteoarthritis, radiculopathy, systemic neurologic conditions)
* Patients having previous injury or surgical treatments of the ankle.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
The Victorian Institute of Sport Assessment-Achilles questionnaire (VISA-A). | 15 minutes
  It consists of eight questions that covered the three domains of pain (questions 1-3), function (questions 4-6), and activity (questions 7 and 8.). Questions one to seven are scored out of 10, and question 8 carries a maximum of 30. Scores are summed to give a total out of 100.

SECONDARY OUTCOMES:
The visual analog scale (VAS). | 15 minutes
  The VAS is a continuous scale consists of a horizontal line (HVAS) usually 10 centimeters (10-100 mm) in length. For pain intensity, the scale is most anchored by no pain (score of 0) and pain as bad as it could be or worst imaginable pain (score of 10

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nasr A. Abdelkader, PhD, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Giza, Egypt